CLINICAL TRIAL: NCT06232733
Title: HELP (HEalthy Lifestyles Project) for Youth With Mental Distress E-Health Intervention: Patient and Healthcare Impacts
Brief Title: HELP (HEalthy Lifestyles Project) for Youth With Mental Distress
Acronym: HELP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Children's Hospital Academic Medical Organization (CHAMO) (Unknown)
Responsible Party: Principal Investigator, Dr. Pat Longmuir, Senior Scientist, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 24
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Mental Health Issue
Keywords: adolescent; healthy lifestyle behavior

STUDY DESIGN:
Intervention Model Description: Immediate or delayed intervention
Who Masked: Outcomes Assessor
Masking Description: It is not possible to blind the participants or families to the study group allocation. Investigators will support delivery of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): Access to HELP e-intervention from 0 to 6 months with kinesiology support.
  Interventions: Behavioral: Healthy Lifestyles Project e-intervention
- Delayed Intervention (Active Comparator): Access to HELP e-intervention from 6 to 12 months with kinesiology support.
  Interventions: Behavioral: Healthy Lifestyles Project e-intervention

INTERVENTIONS:
Behavioral: Healthy Lifestyles Project e-intervention — Virtual lifestyle behaviour change support.
  Other Names: HELP

SUMMARY:
The goal of this clinical trial is to learn about how healthcare providers can support youths' mental health. The main question[s] it aims to answer are:

* Do youth (12 to 17 years of age) who engage in the 6-month HELP e-intervention have a larger improvement in emotional health (measured by the Strengths and Difficulties Questionnaire) than youth who do not receive the intervention?
* Does engagement in the HELP e-intervention improve lifestyle behaviour (physical activity, sleep or screen time)?
* Do youth who engage in the 6-month HELP e-intervention utilize fewer mental healthcare resources, during and for 1 year following study participation, than youth who do not receive the intervention? Participants will receive the HELP intervention for 6 months, either immediately or after waiting 6 months from study enrollment. At 0, 3, 6, and 12 months, participants will answer a series of questionnaires to assess their emotional health and lifestyle behaviors. Researchers will compare the emotional health and lifestyle behaviors of youth who received HELP immediately to those who wait for 6 months prior to the intervention to see if their emotional health or lifestyle behaviors differ.

DETAILED DESCRIPTION:
This study will evaluate the efficacy of 6 months of HELP e-intervention access with kinesiologist support in a randomized controlled trial to determine if the changes in emotional health (primary outcome) and lifestyle behaviors (secondary outcomes) differ from changes among youth with delayed intervention access (control condition). Sustainability of the intervention will be assessed for an additional 6 months. Participants will be youth 12-17 years of age who contact youth mental health services. The unique HELP e-resources developed by the research team utilize age-appropriate graphics and interactive formats developed collaboratively with youth/parent/clinician partners. There are 4 sections: 1) Know Your Habits, 2) Physical Activity, 3) Screen Time, 4) Sleep. A kinesiologist will support participants in the intervention. Study assessments will be completed by researchers blind to study group allocation. Researchers will also evaluate the impact of the HELP e-intervention on the use of mental healthcare services, the need for mental health professional support of lifestyle behaviors and the association between self-reported and objectively measured lifestyle behaviors. It is hypothesized that youth engaging in the HELP e-intervention will have improved emotional health and enhanced lifestyle behaviors in comparison to those receiving the delayed (post 6-months) intervention. It is also hypothesized that changes during the intervention will be maintained for an additional 6 months, and that self-reported measures will accurately reflect objective measurements. Finally, it is hypothesized that youth engaging in the HELP e-intervention will require fewer youth mental health supports, and when supported will be less likely to require treatment directed at lifestyle behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Youth 12-17 years of age seeking, waiting for or receiving support for emotional distress.
* Able to provide informed consent to study participation.
* Able to engage in the HELP e-intervention in English (French translation of the e-modules will not be available until intervention efficacy is established).
* Willing to be randomized to a study group.
* Willing to complete objective behaviour measures if selected (1 of 3 participants).
* Willing to complete the study questionnaires.
* Willing to provide consent for evaluation of mental healthcare system outcomes via their health record.

Exclusion Criteria:

* Identified or suspected eating disorder
* Youth whose health or family status is deemed to be inappropriate for the study as per their most responsible clinician.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire | 6 months
  Youth emotional distress. Minimum score 0. Maximum Score 50. Higher score is lower emotional health.

SECONDARY OUTCOMES:
Habitual Activity Estimation Scale | 6 months
  Self-reported daily physical activity. Minutes and proportion of day spent inactive, somewhat inactive, somewhat active and active for weekend and week days.
Adolescent Sleep Hygiene Scale | 6 months
  Self-reported sleep habits. Minimum score 33. Maximum score 198. Higher score is better sleep hygiene.
Adolescent Sedentary Activity Questionnaire | 6 months
  Self-reported screen time (hours and minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Clare Gray, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Patel R, Longmuir PE, Robb M, Baechler N, Courtney K, Norris M, Goldfield G, Cooligan F, Watson S, Cloutier P, Gray C. Evaluation of the novel HEalthy Lifestyle Project (HELP) youth mental health e-intervention for lifestyle behaviour change and mental healthcare system impact: A randomized controlled trial protocol. PLoS One. 2025 Nov 3;20(11):e0332363. doi: 10.1371/journal.pone.0332363. eCollection 2025. PMID 41183018